CLINICAL TRIAL: NCT07136935
Title: A Multicenter Observational Study of an Integrated Traditional Chinese and Western Medicine Care Model in Post-Acute Treatment of Frail Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC2-105
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Frail Elderly Patients
Keywords: frailty; Chinese and Western Integrated medicine
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): 1. Oral Chinese herbal medicine or decoction
  2. Acupuncture or laser acupuncture treatment
  3. Acupoint massage
  4. Traditional Chinese Medicine Cake Acupoint Application
  5. Nursing and health education and guidance
  6. Dietary hygiene education
  7. Lifestyle health education and sports rehabilitation
  Interventions: Drug: Traditional Chinese Medicine treatment

INTERVENTIONS:
Drug: Traditional Chinese Medicine treatment — 1. Oral Chinese herbal medicine or decoction: prescribe Chinese medicine based on syndrome differentiation and treatment of the patient's condition.
  2. Acupuncture or laser acupuncture treatment: Traditional Chinese medicine practitioners select acupuncture points to treat based on the patient's condition, and treat them once a week.
  3. Acupoint massage: Select treatment acupoints and techniques according to the patient's condition, 20 minutes at a time.
  4. Traditional Chinese Medicine Cake Acupoint Application: Warm Navel Cream to the CV-4 (Guanyuan) acupoint, the application time is 2 to 4 hours.
  5. Nursing and health education and guidance.
  6. Dietary hygiene education: personalized western nutrition and TCM dietary guidance suggestions based on TCM constitution syndromes.
  7. Lifestyle health education and sports rehabilitation: Playing Baduanjin, ten skilled hand exercise, and health preservation videos, and providing personalized TCM exercise recommendations.

SUMMARY:
Exploring the Impact and Effectiveness of an Integrated Traditional Chinese and Western Medicine Treatment Model in Post-Acute Care for Frail Older Patients.

DETAILED DESCRIPTION:
Frailty Syndrome is a common syndrome in the geriatric population, with prevalence of 14% in a population of 65 years old and 26% in 85 years old. Clinically, frailty syndrome is associated with increased vulnerability, decreased physical strength and a decline in daily function. There are five main signs include low grip strength, low energy, slowed walking speed, low physical activity, and/or unintentional weight loss. Patients with frailty syndrome are more likely to experience adverse events such as falls, fractures, hospitalizations, and infections, which may even lead to increased mortality. The progression of frailty can significantly reduce patients' quality of life, and increase the medical burden along with burden on families and society.In the modern society as people live longer lives, the incidence of frailty syndrome is increasing year by year, and strategies for managing and delaying the frailty syndrome progression are warranted.

Traditional Chinese Medicine (TCM) is based on empirical clinical experience over thousands of years and long-established knowledge. It implements "syndrome differentiations" that are based on regulating the balance of Qi (energy) and blood in the body, restoring organ functions, and improving the body's self-regulation ability, through those concepts TCM provides a treatment potential. For frailty syndrome, TCM can play an important role in improving patients' physical strength, enhancing muscle strength, alleviating chronic inflammation, and improving quality of life.TCM has the advantages of simplicity, safety, and is suitable for the elderly. Therefore, the comprehensive treatment model of TCM not only provides a potentially effective intervention method for patients with frailty syndrome but also provides new approaches for the integrative management of geriatric diseases.

Methods: patients with mild to moderate frailty syndrome will be included in this study. Western physicians and Chinese medicine practitioners jointly evaluate those who are suitable for inclusion. The combined Chinese and Western medicine intervention will begin after informed consent signature by patients or their families. TCM interventions include acupuncture, herbal medicine/ herbal formulas, acupoint stimulation, TCM diet and lifestyle education, etc. The TCM doctor will determine the type of TCM intervention recommended based on the patient's needs and TCM diagnosis and discussion with Western medicine doctor. A total of 20 patients are expected to be admitted and case records will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients aged ≥75 years.
2. A history of at least one of the following conditions: Parkinson's disease, chronic obstructive pulmonary disease (COPD), mild dementia, or chronic kidney disease at stage 3 or above.
3. Hospitalized due to an acute illness (length of hospital stay >72 hours).
4. Functional decline within one month after completion of treatment.
5. Clinical Frailty Scale (CFS) score of 5-7 (indicating moderate or greater frailty, with retained rehabilitation potential).
6. Can answer clinical questionnaires and scales.

Exclusion Criteria:

1. Medically unstable (requiring intensive medical interventions, diagnostic testing, or supplemental oxygen).
2. Unable to cooperate with treatment or communication.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Study of Osteoporotic Fractures | At baseline, End of treatment(4 weeks)
  Measured by the Study of Osteoporotic Fractures (SOF Index) ,score of 0~2 : 0=robust,1 =prefrail,2= frail.
comprehensive geriatric assessment | At baseline, End of treatment(4 weeks)
  Measured by comprehensive geriatric assessment(CGA)
Body Constitution Questionnaire / Constitution in Chinese Medicine Questionnaire | At baseline, End of treatment(4 weeks)
  Measured by Body Constitution Questionnaire(BCQ) / Constitution in Chinese Medicine Questionnaire(CCMQ)

SECONDARY OUTCOMES:
Height | At baseline, End of treatment(4 weeks)
  height in cm.
Weight | At baseline, End of treatment(4 weeks)
  weight in kilograms
Calf circumference | At baseline, End of treatment(4 weeks)
  Keep your knee bent at a 90-degree angle, and measure the circumference of your calf at its widest point horizontally.
Grip strength | At baseline, End of treatment(4 weeks)
  Use a handheld Jamar dynamometer in a sitting position with the elbow bent 90-degrees ,You can use either hand or your dominant hand. Record the highest value from two measurements.
Gait speed | At baseline, End of treatment(4 weeks)
  6-m usual walking speed test

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan